CLINICAL TRIAL: NCT00717145
Title: Food Effects on the Relative Bioavailability of a Risedronate 20 mg Delayed-release [DR] Tablet and to Compare the 20 mg DR Tablet to 35 mg DR and 35 mg Immediate-release Tablets
Brief Title: Food Effects on the Relative Bioavailability of Different Dosages of Risedronate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2008052
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Postmenopausal; Non-lactating; Surgically Sterile
Keywords: bioequivalence
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): One risedronate 20 mg DR tablet taken following an overnight fast, followed by a 4-hour fast.
  Interventions: Drug: risedronate
- 2 (Experimental): One risedronate 20 mg DR tablet taken following an overnight fast, within 5 minutes after ingesting a high-fat meal; no additional food will be allowed for at least 4 hours post-dose.
  Interventions: Drug: risedronate
- 3 (Experimental): One risedronate 35 mg DR tablet taken following an overnight fast, within 5 minutes after ingesting a high-fat meal; no additional food will be allowed for at least 4 hours post-dose.
  Interventions: Drug: risedronate
- 4 (Experimental): One risedronate 35 mg IR tablet taken following an overnight fast, 30 minutes before ingesting a high-fat meal; no additional food will be allowed for at least 4 hours post-dose.
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — one risedronate 20 mg DR tablet
  Arms: 1
Drug: risedronate — One risedronate 20 mg DR tablet
  Arms: 2
Drug: risedronate — One risedronate 35 mg DR tablet
  Arms: 3
Drug: risedronate — One risedronate 35 mg IR tablet
  Arms: 4

SUMMARY:
Randomized, open-label, multi-center, 4-treatment, 4-period crossover study. The study will consist of a screening visit, study center admission (preceding Treatment Periods 1, 2, 3, and 4), 4 treatment periods (4 days each), 3 washout periods (14 to 17 days in duration separating each treatment period), and exit procedures.

ELIGIBILITY:
Inclusion Criteria:

* non-lactating and either surgically sterile or postmenopausal:
* body mass index less than or equal to 32 kg/m2 at screening

Exclusion Criteria:

* No use of a bisphosphonate within 1 month
* no history of GI disease
* no use of any medications within 7-14 days prior to scheduled dosing day

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Assess the relative bioavailability of the risedronate 20 mg DR tablet administered immediately after a high-fat meal compared to the risedronate 35 mg IR tablet administered 30 minutes prior to a high-fat meal. | 4 Days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Gainesville, Florida
  - Research site, Miramar, Florida
  - Research Site, Austin, Texas